CLINICAL TRIAL: NCT02580617
Title: A Phase 1 Clinical Study to Evaluate the Safety of Allogeneic Adipose-derived Stem Cells in the Subjects With Crohn's Disease
Brief Title: A Study to Evaluate the Safety of ALLO-ASC-CD for Treatment of Crohn's Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-ASC-CD-101
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALLO-ASC (Experimental): Group 1: 5.0 x 10^7 cells Group 2: 7.5 x 10^7 cells Group 3: 10.0 x 10^7 cells
  Interventions: Biological: ALLO-ASC

INTERVENTIONS:
Biological: ALLO-ASC — Infusion for Crohn's disease
  Other Names: ALLO-ASC-CD

SUMMARY:
This is a phase I study to evaluate the safety of ALLO-ASC-CD for the treatment of crohn' disease. ALLO-ASC-CD is intravenous infusion containing allogenic adipose-derived mesenchymal stem cells.

DETAILED DESCRIPTION:
Adipose-derived stem cells are directed to injured tissue, and reduce inflammation. Furthermore, their immunomodulatory effects are significant for treating immune-related diseases, such as crohn's disease. Finally, ALLO-ASC-CD may provide a new option in treating a crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 to 65 years of age
2. Subject who is diagnosed Crohn's disease by endoscopic or radiologic result during more than 6 months
3. Subject who show intolerance or failure of conventional therapy (steroids, immunosuppressive and TNF-alpha inhibitor)
4. Subject who is included CDAI 220-450 during screening period
5. CRP>0.5mg/dL during screening period
6. Subject who show affected sites by crohn's disease in either ileum and large intestine or both of them, including more than 1 nonanastomotic ulcers as a result of colonoscopy.
7. Subjects who satisfy those clinical examination value below during screening period.

   A. Hemoglobin ≥ 8.0g/dL B. WBC ≥ 3,000/μL C. Lymphocyte ≥ 500/μL D.100,000/μL ≤ Platelet ≤ 1,200,000/μL E. AST and ALT ≤ 3 x the upper limit of normal F. ALP ≤ 3 x the upper limit of normal G.Serum creatinine ≤ the upper limit of normal H.Serum albumin ≥ 2.0g/dL I.PT , aPTT≤ the upper limit of normal
8. Negative for urine beta-HCG for women of childbearing age.
9. Subject is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Subject with gastro-intestinal tract A. Crohn's disease which is invaded only proximal ileum. B. The evidence of an intra abdominal abscess during screening period. C. The evidence of an abscess around the anus during screening period. D. Conditions of subtotal colectomy or total colectomy. E. Short bowel syndrome. F. Subject who conduct elemental diet, tube feeding or parenteral nutrition within 3 weeks before enrollment.

   G. Subject who have ileostomy or colostomy. H Subject who have a bowel stricture of large intestine that may be significant by PI's decision during screening period.

   I. In case that the PI anticipates that patients need to get a surgical intestinal tract surgery caused by crohn's disease.

   J. Subject who have adenoma of large intestine K. Subject who have chronic inflammation-associated dysplasia.
2. Subjects who have been received biological therapy within 60 days of enrollment..
3. Subject with infectious disease A. Acute or chronic active HBV, HAV and HIV B. Active tuberculosis. C. IGRA (Interferon-Gamma Release Assay) positive D. All kinds of live vaccine inoculation except influenza vaccine within 4weeks before registration E. Pneumonia, pyelonephritis and Infection of Clostridium within 4weeks during screening visit.

   F.Subject has history of bacteremia or other serious bacterial or fungal infection in past 3 months.
4. Subject who has malignant tumor or which is not cured yet
5. Subject has any serious disease, in the opinion of the Investigator, would interfere with the evaluation of the study.
6. Subject who has history of blood clots and other pathological arterial thrombosis or venous thrombosis
7. Subject who has a hypersensitive reaction to bovine-derived proteins
8. Subject who is surgery or trauma within 6 weeks before registration
9. Subject who is pregnant or breast-feeding.
10. Subjects who are unwilling to use an "effective" method of contraception during the study
11. Subject who is experienced stem cell therapy
12. Subject who has been enrolled in another clinical study within 4weeks days of screening
13. Subject who has history of alcohol or drug abuse.
14. Subject who is not able to understand the objective of this study or to comply with the study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2015-11-09 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety (Clinically measured abnormality of laboratory tests and adverse events) | up to 4 weeks
  Clinically measured abnormality of laboratory tests and adverse events

SECONDARY OUTCOMES:
CDAI value | up to 4 weeks
  Change in the CDAI value
The ratio of patients applicable to CDAI <150 | Week 4
  The ratio of patients applicable to CDAI <150

CONTACTS AND LOCATIONS:
Overall Officials: Won Ho Kim, Principal Investigator — Yonsei University
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea